CLINICAL TRIAL: NCT04180475
Title: Adherence to Medical Treatments for Telemedicine Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed due to not able to find any real stroke patients interested to participate.
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, John A Stankovic, Professor, Comp Science, University of Virginia
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 21012
Record Dates: First submitted 2019-10-30; First posted 2019-11-27 (Actual); Results first posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-02

CONDITIONS: Stroke; Medication Adherence
Keywords: Remote monitoring
MeSH Terms: conditions — Stroke; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Phase 1 - determine the feasibility of the Apple Watch medication/exercise reminder system MedRem by deploying the system to control subjects.
  Phase 2 of study- assess the subjects' adherence to medications, exercise and checking heart rate (and quality of the exercise), with the use of MedRem
  • assess the acceptance and usability of the MedRem system.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- MedRem application (Experimental): MedRem smartwatch application
  Interventions: Device: MedRem application

INTERVENTIONS:
Device: MedRem application — Medication adherence smartwatch application

SUMMARY:
This study will test the feasibility of MedRem, a novel medication reminder and tracking system on wearable wrist devices, specifically with the Apple Watch 4. The study team will load the MedRem app onto two Apple Watch 4s for use during the study. As the device is placed on the wrist, it is free from the limitations of smartphones. However, one of the major challenges in developing interactive systems for wrist devices is their form factor. The touch screens available on these devices are tiny and much smaller compared to smart phones and tablet computers. MedRem enables user interactions by incorporating speech recognition and text-to-speech features along with clever interface design. The tiny display of the device is used for minimal inputs and outputs, while a user can retrieve and provide more information from/to the system through voice commands. Personalized models are built and updated over time to reduce errors in recognizing users' voice commands, and thus better user experience is provided.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1 (Controls)

  * 18 - 75 years old
  * Good general health (self-reported), with no history of cerebral vascular accident (CVA)
  * English-speaking
  * Willingness and ability to comply with scheduled visits and study procedures

Phase 2 (Stroke Patients)

* 18 - 75 years old
* English-speaking
* Willingness and ability to comply with scheduled visits and study procedures
* Have requirements for home- based therapy regimens (i.e. physical/occupational therapy)
* Require medications for secondary stroke prevention (e.g. antithrombotic therapy to prevent ischemic stroke, stroke risk factor management with blood pressure, diabetes, cholesterol medications).
* Have a Modified Rankin Scale for Neurologic Disability (MDS) of 2 - 4

Exclusion Criteria:

* Phase 1 (Controls)

  * Pregnant women, fetuses, neonates, children, prisoners, cognitively impaired, non-English speaking subjects
  * Prohibitive cognitive impairments or language deficits
  * Does not have wireless internet connection at home

Phase 2 (Stroke Patients)

* Pregnant women, fetuses, neonates, children, prisoners, cognitively impaired, non-English speaking subjects
* Have a Modified Rankin Scale for Neurologic Disability (MDS) of 0-1 or 5
* Prohibitive cognitive impairments or language deficits
* Significant weakness, dystonia, or spasticity that will prevent proper use and response to the Apple Watch device
* Live in nursing home or rehabilitation facility
* Does not have wireless internet connection at home

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Stankovic, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MedRem Application
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MedRem Application
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Use of MedRem System
Description: Assess the patients' adherence to medications and exercise. Adherence will be measured by patient responses to questions prompted by the MedRem System.
Time Frame: 30 days
Population: No data were collected for this Outcome Measure
Arm/Group | MedRem Application
Number analyzed (Participants) | 0

2. Primary Outcome: Assessment of Survey
Description: Acceptance and usability will be measured by the Intervention Patient MedRem Usability Survey. Steps were taken and distance covered data will also be collected from the Apple Watch.
Time Frame: 30 days
Population: No data were collected for this Outcome Measure
Arm/Group | MedRem Application
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: End of Week 1
Arm/Group | MedRem Application
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT04180475/Prot_SAP_000.pdf